CLINICAL TRIAL: NCT04609527
Title: Management of Placenta Accreta Spectrum
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Osama Saber Thabet Abdalmageed, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Placenta Accreta
Record Dates: First submitted 2020-10-15; First posted 2020-10-30 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Placenta Previa; Placenta Accreta
Keywords: placenta; accreta; praevia; hyterectomy; PPH
MeSH Terms: conditions — Placenta Previa; Placenta Accreta

STUDY DESIGN:
Intervention Model Description: All women with placenta praevia and previous scar in the uterus. Surgical management and follow up will be defined
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Management of placenta accreta spectrum — Conservative and radical (hysterectomy) treatment of placenta accreta. Follow up to the patients to detect the impact of treatment imposed A novel technique which early identification and repait of uterine wall defects resulted from invasion of the uterine wall by the placenta.

SUMMARY:
placenta accreta spectrum is group of disorders which have a depate about the best way of management. this is a descriptive study about the best techniques to reduce morbidity and mortalities related to it.

DETAILED DESCRIPTION:
placenta accreta spectrum is group of disorders which have a depate about the best way of management. this is a descriptive study about the best techniques to reduce morbidity and mortalities related to it.

1. surgical management of placenta accreta
2. short term follow up to the outcomes
3. long term follow up

ELIGIBILITY:
Inclusion Criteria:

* All placenta accreta e high possibility of placenta accrete
* consent
* easy follow up visits

Exclusion Criteria:

* bleeding tendency
* associated medical disorder hypertension, diabetes, preeclapsia..

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Failure of the novel conservative management | 3 hours
  Need to do peripartum hysterectomy or patient death
Estimated amount of blood loss | 6 hours
  The estimated amount of blood loss during and after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Osama Abdalmageed, Asyut, Non-US/Non-Canadian
  - Assiut University, Asyut

IPD SHARING:
Plan to Share IPD: Undecided